CLINICAL TRIAL: NCT01235286
Title: Effects of Remote Ischemic Preconditioning in Cutaneous Microcirculation of Anterolateral Thigh Flaps
Brief Title: Cutaneous Remote Ischemic Preconditioning in Plastic Surgery
Acronym: RIPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Robert Kraemer, Hannover Medical School, Plastic, Hand and Reconstructive Surgery
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: Kraemer001
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: Ischemic Preconditioning
Keywords: remote ischemic preconditioning, free flap, microcirculation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- remote ischemic preconditioning (Experimental)
  Interventions: Procedure: remote ischemic preconditioning

INTERVENTIONS:
Procedure: remote ischemic preconditioning — A standardized location for microcirculatory assessment was determined on the left leg of each participant between the proximal and distal third of a drawn line between the anterior superior iliac spine and the lateral aspect of the Patella.
  The healthy subjects had to rest before starting data assessment in a horizontal position for 15 minutes. The probe was taped on the left upper leg in a standardized manner after localizing the measuring point. A blood pressure cuff was applied on the contralateral upper arm. Baseline data was assessed over 5 minutes before starting remote ischemia. Three circles of a five minute ischemia were applied at the contralateral right upper arm at suprasystolic levels. Parameters of microcirculation were assessed continuously over time. Microcirculation during the reperfusion phase was ascertained over 10 minutes after first and second remote ischemia and 15 minutes after the third remote ischemia.

SUMMARY:
Background: In plastic and reconstructive surgery, free flaps are routinely used for treatment of soft tissue defects. Treatment strategies aim at reducing or preventing flap necrosis by conditioning tissue tolerance against ischemia. Although previous studies indicate that remote ischemic preconditioning (RIPC) is a systemic phenomenon, only a few studies have focused on the elucidation of its mechanisms of action. Therefore, the aim of this study is to evaluate the microcirculatory effects of remote ischemic preconditioning on a potential free flap location in a human in-vivo setting for the first time.

Conclusion: Remote ischemic preconditioning improves cutaneous tissue oxygen saturation, arterial capillary blood flow and postcapillary venous flow in a remote free flap donor location. To what extent remote preconditioning might ameliorate the reperfusion injury of free flap transplantation, further clinical trials have to evaluate both in the means of microcirculatory assessment and partial or total flap loss as end points of these studies.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female subjects aged 18 to 35 years

Exclusion Criteria:

* soft tissue inflammation or osteomyelitis, peripheral arterial occlusive disease, vasculitis, chronic kidney or liver disease, cardiac dysfunction, arterial hypotension and any type of vasoactive medication, i.e. ß-blockers, calcium channel blockers, nitroglycerin

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in microcirculation
  * capillary blood flow [arbitrary units AU]
  * capillary blood velocity [AU]
  * tissue oxygen saturation [%]
  * relative postcapillary venous filling pressure [AU]

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kraemer, MD, Principal Investigator — Medical School Hannover, Plastic, Hand and Reconstructive Surgery
Locations (1):
- Medical School Hannover, Hanover, Germany

REFERENCES:
- [Derived] Kraemer R, Lorenzen J, Kabbani M, Herold C, Busche M, Vogt PM, Knobloch K. Acute effects of remote ischemic preconditioning on cutaneous microcirculation--a controlled prospective cohort study. BMC Surg. 2011 Nov 23;11:32. doi: 10.1186/1471-2482-11-32. PMID 22111972